CLINICAL TRIAL: NCT02667795
Title: Improving Physical Fitness Prior to Colorectal Surgery: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SNE 2447
Record Dates: First submitted 2016-01-07; First posted 2016-01-29 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Bowel Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitored walking based exercise (Experimental): Participants will be given a personalised daily exercise target. Participants will be given an activity tracker (a Fitbit ZipTM). The participants will be asked to wear the device all day to monitor their activity. Once a day the participants will be asked to complete the walking target they have been given at completion of their baseline assessment. This target should be completed in one go. The walking programme will last a minimum of 2 weeks and a maximum duration of 4 weeks. The length of time will depend on the length of time between recruitment and when the participant is scheduled to have their surgery.
  Interventions: Other: Monitored walking based exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Monitored walking based exercise — Monitored walking based exercise
  Arms: Monitored walking based exercise

SUMMARY:
It is generally accepted that physically fit patients cope much better with the stress of surgery and recover faster. Consequently several research studies have tried to increase people's level of fitness before they have surgery. These previous research studies have usually required patients to carry out intense, structured exercise programmes that involve going to a gym. However such programmes are not 'user friendly' especially if people are not used to taking a lot of exercise. In this pilot study we want to test the feasibility of a home based programme that tries to increase patients' level of fitness by gradually increasing the number of steps they walk every day.

DETAILED DESCRIPTION:
Participants will be randomised into one of two groups. One group of participants will be asked to increase their level of activity by gradually walking further (the exercise group) and the other group will carry on with their usual level of activity (the usual activity group) .

Assessments People in both groups will have an assessment on 3 occasions: when they join the study, just before surgery and 3 months after surgery.

This assessment involves:

Walking for 6 minutes up and down a corridor to see how far they can walk. Asking them for some information about their medical history Completing three questionnaires about how they are feeling and their quality of life.

People who are randomised to the exercise group will be advised about how many steps to take based on how they did in the initial walking assessment. The number of days or weeks they will be asked to take a daily walk will depend on how much time there is between them joining the study and the date of their surgery. We think this will be about 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Requiring elective resectional bowel surgery
* Gives consent to participate in the study

Exclusion Criteria:

* Younger than 18 years of age.
* A history of unstable angina/unstable coronary artery disease or a heart attack in the previous month.
* Any heart related disease including but not limited to aortic stenosis, pericarditis or any thromboembolic disease.
* Severe Infections and fever.
* Uncontrolled metabolic diseases.
* Resting heart rate of more than 120 BPM.
* Systolic blood pressure of more than 180 mm Hg or diastolic blood pressure of more than 110 mm Hg.
* Recent cerebrovascular accident.
* Pregnancy
* Pre-existing severe physical disability.
* Unwilling to allow their GP to be informed of their participation in the study.
* Not able or unwilling to consent to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Change in fitness as assessed by Six Minute Walk Test | Will be done at recruitment, prior to surgery and 3 months post operatively
  Fitness assessment

SECONDARY OUTCOMES:
The EQ-5D | Will be done at recruitment, prior to surgery and 3 months post operatively
  Quality of life assessment
EORTC QLC-C30 | Will be done at recruitment, prior to surgery and 3 months post operatively
  Quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: John Macfie, MBChB, MD, Study Director — York Teaching Hospitals NHS Foundation Trust
Locations (1):
- Scarborough General Hospital, Scarborough, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No